CLINICAL TRIAL: NCT03217383
Title: Predictive Accuracy of MATRx Plus in Identifying Favorable Candidates for Oral Appliance Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zephyr Sleep Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZCP201703
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Sleep Apnea; Sleep Apnea, Obstructive; Sleep Disordered Breathing
Keywords: Oral appliance therapy; mandibular protrusion
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Masking Description: Though the study only has one study arm, the participant, medical PI, dental PI will be blinded to the test prediction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MATRx plus test (Experimental): All study participants will receive the same test protocol. All participants will complete the MATRx plus theragnostic test and receive a prediction of oral appliance outcome. All participants will then receive a custom oral appliance set to the predicted protrusive position or a sham position, and outcome home sleep tests will be performed with the custom oral appliance in place to determine if the test prediction was correct.
  Interventions: Device: MATRx plus

INTERVENTIONS:
Device: MATRx plus — The MATRx plus test is a 2- or 3-night home sleep test that uses temporary titration trays to move the lower jaw in response to respiratory events. The purpose of the test is to predict oral appliance therapy outcome, and to provide a protrusive position for individuals predicted to experience therapeutic success.

SUMMARY:
Obstructive sleep apnea (OSA) is a common disease that is largely un-diagnosed and untreated. Standard treatment for obstructive sleep apnea, nasal continuous positive airway pressure (CPAP), entails use of a nose mask to deliver positive pressure which dilates the pharynx and eliminates obstruction. This therapy is highly efficacious and benign but is associated with low adherence, particularly in non-sleepy apneics with disease of mild and moderate severity. The principal alternative to CPAP therapy is oral appliance (OA) therapy in which a custom made mandibular advancement splint (MAS) is used to protrude the mandible during sleep, thereby opening the pharyngeal airway. OA therapy, while preferred and well accepted by most participants, is not uniformly efficacious. Additionally, uncertainty regarding the patient's response to OAT and the effective target mandibular position can lead to a significant time span between diagnosis and initiation of effective treatment. Furthermore, knowledge of the effective target mandibular position supports the use of new OA design and manufacturing processes that can further reduce the time and cost in delivering the therapy.

Zephyr Sleep Technologies (the Sponsor) has developed a method of identifying OAT responsive participants and their efficacious mandibular protrusion. Recently, Zephyr Sleep Technologies developed a portable device that avoids this requirement and can be used in a multi-night test in the home. Using a feedback controlled mandibular positioner (FCMP), the device measures and analyzes respiratory airflow and oxygen saturation and makes decisions in real-time about moving the mandible. The FCMP device was tested in a blinded, bi-phase clinical study in which participants with mild-to-severe sleep apnea (n=202) underwent two full-night studies in the home. Data from phase 1 were used to develop a predictive method, and data from phase 2 were used to prospectively test the accuracy of the predictive method. An efficacious mandibular position was also predicted, and each participant was treated with a custom oral appliance set to that position. Data from both phases were used to evaluate the feasibility of use of the device in the home.

A random forest machine learning system was used to develop and test the predictive method. The overall oral appliance success rate was 76% for phase 1 and 71% for phase 2. The overall predictive accuracy was 88%. Values for sensitivity and specificity were 85% and 93%, respectively. Positive and negative predictive values were 97% and 72%, respectively. The effective target protrusive position was identified in 86% of cases. The studies were conducted independently by the participants in their homes, though due to limitations in the early prototype design, a clinical coordinator visited the home to set up the equipment prior to each night of study. No significant problems were encountered, and no significant risks were identified. The results of the clinical trial show that the auto-titrating mandibular positioner is suitable for use in the home and accurately predicts OAT outcome as well as target protrusive position.

Based on the results of this study, Zephyr developed a commercially available device which has been approved for sale in Canada (Health Canada device license #97614). The device, branded MATRx plus, functions as both a sleep recorder as well as a home-based system to select patients for oral appliance therapy. This commercially available device is currently being used in three separate usability trials to quantify the usability of the device and the benefits of an improved workflow through adoption of the new technology in a dental practice.

Evidence has recently appeared to indicate that the change in pharyngeal volume caused by protrusion of the mandible, measured while awake, correlates with the change in apnea-hypopnea index (AHI) achieved by OAT, measured while asleep. This is the first convincing evidence that an awake measurement of the pharyngeal airway correlates with the improvement in respiratory status during sleep induced by an oral appliance. The implication is that a simple conebeam CT of the pharynx can predict outcome with OAT. Accordingly, we shall carry out conebeam CTs in the research protocol, both at rest position of the mandible and at 90% of maximal protrusion.

The purpose of this study is to test whether the predictive accuracy of the FCMP in the home environment is improved by the commercial design and whether patients predicted to be suitable for oral appliance therapy have long term adherence.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common disease that is largely un-diagnosed and untreated. Standard treatment for obstructive sleep apnea, nasal continuous positive airway pressure (CPAP), entails use of a nose mask to deliver positive pressure which dilates the pharynx and eliminates obstruction. This therapy is highly efficacious and benign but is associated with low adherence, particularly in non-sleepy apneics with disease of mild and moderate severity. The principal alternative to CPAP therapy is oral appliance (OA) therapy in which a custom made mandibular advancement splint (MAS) is used to protrude the mandible during sleep, thereby opening the pharyngeal airway. OA therapy, while preferred and well accepted by most participants, is not uniformly efficacious. Additionally, uncertainty regarding the patient's response to OAT and the effective target mandibular position can lead to a significant time span between diagnosis and initiation of effective treatment. Furthermore, knowledge of the effective target mandibular position supports the use of new OA design and manufacturing processes that can further reduce the time and cost in delivering the therapy.

Zephyr Sleep Technologies (the Sponsor) has developed a method of identifying OAT responsive participants and their efficacious mandibular protrusion. A remotely controlled mandibular positioner (RCMP) is used during polysomnographic monitoring to vary the mandibular position. The in-lab version of the device, requiring use of a sleep technologist during a polysomnographic study, was shown to accurately predict outcome with a custom oral appliance in a triple-blind, prospective, predictive study in sixty-seven participants with mild-to-severe sleep apnea (specificity: 92%; PPV: 94%; sensitivity: 86%; NPV: 83%). In addition, the predicted target mandibular protrusive position proved efficacious in 87.5% of cases. While accurate in prospectively identifying oral appliance responders, the availability and utility of the RCMP device is limited by the requirement of a polysomnographic study.

Recently, Zephyr Sleep Technologies developed a portable device that avoids this requirement and can be used in a multi-night test in the home. Using a feedback controlled mandibular positioner (FCMP), the device measures and analyzes respiratory airflow and oxygen saturation and makes decisions in real-time about moving the mandible. The FCMP device was tested in a blinded, bi-phase clinical study in which participants with mild-to-severe sleep apnea (n=202) underwent two full-night studies in the home. Data from phase 1 were used to develop a predictive method, and data from phase 2 were used to prospectively test the accuracy of the predictive method. An efficacious mandibular position was also predicted, and each participant was treated with a custom oral appliance set to that position. Data from both phases were used to evaluate the feasibility of use of the device in the home.

A random forest machine learning system was used to develop and test the predictive method. The overall oral appliance success rate was 76% for phase 1 and 71% for phase 2. The overall predictive accuracy was 88%. Values for sensitivity and specificity were 85% and 93%, respectively. Positive and negative predictive values were 97% and 72%, respectively. The effective target protrusive position was identified in 86% of cases. The studies were conducted independently by the participants in their homes, though due to limitations in the early prototype design, a clinical coordinator visited the home to set up the equipment prior to each night of study. No significant problems were encountered, and no significant risks were identified. The results of the clinical trial show that the auto-titrating mandibular positioner is suitable for use in the home and accurately predicts OAT outcome as well as target protrusive position.

Based on the results of this study, Zephyr developed a commercially available device which has been approved for sale in Canada (Health Canada device license #97614). The device, branded MATRx plus, functions as both a sleep recorder as well as a home-based system to select patients for oral appliance therapy. This commercially available device is currently being used in three separate usability trials to quantify the usability of the device and the benefits of an improved workflow through adoption of the new technology in a dental practice.

ProSomnus Sleep Technologies has developed a digitally designed and milled sleep appliance called the MicrO2. This device is designed to accurately represent the bite and targeted mandibular position, minimize tongue interference, maintain the targeted mandibular position throughout the night using 90-degree fin angles and use a novel titration process that can reduce error in patient/doctor titration position selection. This device coupled with a digital workflow and outcome of the FCMP is postulated to provide an increase in efficiency of delivering efficacious treatment to the patient from diagnosis to final therapy.

Evidence has recently appeared to indicate that the change in velo-pharyngeal volume caused by protrusion of the mandible, measured while awake, correlates with the change in apnea-hypopnea index (AHI) achieved by OAT, measured while asleep. This is the first convincing evidence that an awake measurement of the pharyngeal airway correlates with the improvement in respiratory status during sleep induced by an oral appliance. The implication is that a simple conebeam CT of the pharynx can predict outcome with OAT. Accordingly, we shall carry out conebeam CTs in the research protocol, both at rest position of the mandible and at 90% of maximal protrusion.

The purpose of this study is to test whether the predictive accuracy of the FCMP in the home environment is improved by the commercial design and whether patients predicted to be suitable for oral appliance therapy have long term adherence.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 21 and 80 years
2. Obstructive sleep apnea (ODI and AHI > 10hr-1)
3. Body mass index less than 45 kg/m2
4. Neck circumference less than 50 cm
5. Absence of severe oxyhemoglobin desaturation during sleep as indicated by a mean value of oxygen saturation (SaO2) greater than 87 percent
6. Mandibular range of motion greater than 5 mm
7. Adequate dentition (10 upper and 10 lower teeth)
8. Ability to understand and provide informed consent
9. Ability and willingness to meet the required schedule

Exclusion Criteria:

1. Inability to breathe comfortably through the nose
2. Central Sleep Apnea (>50% of apneas are central)
3. Anticipated change in medical therapy that could alter the severity of OSA during the protocol
4. Anticipated change in body weight (5% or more) during the protocol
5. Symptomatic, non-respiratory sleep disorder, e.g., restless leg syndrome or chronic insomnia
6. Severe respiratory disorder(s) other than sleep disordered breathing
7. Loose teeth, faulty restorations, or advanced periodontal disease
8. Participation in other studies that could interfere with study protocol
9. Pregnant or nursing
10. Patients with heart failure
11. Cerebral vascular incident within the last 12 months
12. Use of pacemaker or other life supporting device
13. Regular use of CPAP or oral appliance therapy within the last 1 month

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
Sensitivity | 6 weeks
  The hypothesis that sensitivity is greater than 0.50 (50%) when the MATRx plus device is used independently by patients in the home will be tested.
Oral appliance compliance | 12 months
  The long-term use of the oral appliance in patients selected for oral appliance therapy by the MATRx plus device will be documented.

SECONDARY OUTCOMES:
Usability | 3 days
  The usability of the MATRx plus device in the home will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: John Remmers, MD, Principal Investigator — Zephyr Sleep Technologies
Locations (1):
- Zephyr Sleep Technologies, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Derived] Mosca EV, Grosse J, Remmers JE. Oral appliance therapy is highly efficacious at reducing sleep apnea-specific hypoxic burden, a metric predictive of cardiovascular morbidity and mortality. J Clin Sleep Med. 2025 Jul 1;21(7):1185-1190. doi: 10.5664/jcsm.11622. PMID 40123555
- [Derived] Mosca EV, Bruehlmann S, Zouboules SM, Chiew AE, Westersund C, Hambrook DA, Jahromi SAZ, Grosse J, Topor ZL, Charkhandeh S, Remmers JE. In-home mandibular repositioning during sleep using MATRx plus predicts outcome and efficacious positioning for oral appliance treatment of obstructive sleep apnea. J Clin Sleep Med. 2022 Mar 1;18(3):911-919. doi: 10.5664/jcsm.9758. PMID 34747691